CLINICAL TRIAL: NCT00725166
Title: Human Muscle Gene Expression Profiles in Young and Old Men
Acronym: CERA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Fondation des Caisses d'Epargne Rhône-Alpes (Unknown); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Clément CAILLAUX, CHU de Saint-Etienne
Other Study IDs: 0708102; 2008-A00374-51
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Elderly; Sarcopenia
Keywords: Aging; Biopsy; Skeletal muscle; Molecular biology; Genetic markers; Gene expression regulation; Young and old men; Healthy volunteers
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, muscle
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young: Young men 19-25 years old
  Interventions: Other: Skeletal muscle aging
- Old: old men 70-76 years old, who participate in the PROOF study (NCT 00759304)
  Interventions: Other: Skeletal muscle aging

INTERVENTIONS:
Other: Skeletal muscle aging — W1 - Blood test
  * Maximal voluntary contraction of quadriceps
  * Hydrostatic weighing
  W2 - Maximal metabolic test using a cycloergometer
  W3 - Muscular biopsy

SUMMARY:
To reach the goals of living longer in better medical conditions, many countries reach the same conclusion: new strategies have to be developed to avoid, or at least limit, the effects of age; this requires a better knowledge of the mechanisms of aging. Our project focuses on the loss of muscle mass associated with aging, called sarcopenia. Sarcopenia unavoidably leads to impaired mobility and poor balance, which contributes to loss of functional autonomy and to increased prevalence for severe falls. Skeletal muscle also plays a central role as a reserve for energy and amino acids. Hence, sarcopenia further triggers severe side metabolic effects such as frailty among elderly persons. The precise mechanisms of muscle aging are still mostly unknown, although many theories have been proposed.

The present study aims at better understanding the mechanisms of skeletal muscle loss associated with aging. Using muscle biopsies from young and old subjects, the differential expression profiles of mRNA will be obtained through chips that will evaluate more than 39000 transcripts. On the same samples, proteomic analyses will involve two complementary approaches: (1) bidimensional electrophoresis (2DGE) coupled to mass spectrometry (MALDI-ToF) for dominant proteins; (2) Western-blot (more than 800 antibodies) targeting regulating proteins not detectable using 2DGE. Complementary histological studies (immunohisto-fluorescence, confocal microscopy) will specify the localisation of the major biomarkers in the muscle biopsies.

The results of that research will have applications in the medium term and will lead to nutritional interventions to modulate specific metabolic pathways and improve the quality of life in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated or beneficiary of a social security category
* Having signed the inform consent form
* Having signed the genetic consent form

Exclusion Criteria:

* Antiaggregant platelet treatment
* Type 2 diabetes
* Body Mass Index > 25
* Severe renal disease
* CRP > 10
* Abnormal clotting test
* Allergies to local anesthetics

Ages: 19 Years to 76 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young : students of the Saint-Etienne's university. Old : men who participate in the PROOF study
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To identify the differential expression profiles (proteomics, transcriptomics) in skeletal muscle between young and old men | During biopsie (W3)

SECONDARY OUTCOMES:
To specify the localisation of the major biomarkers in the muscle biopsies. | During biopsie (W3)
To compare muscular energy metabolic enzymatic activities between young and old men | during biopsie (W3)
To compare the number of muscular stem cells between young and old men | during biopsie (W3)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel BECHET, PhD, Study Chair — INRA Clermont-Ferrand; Jean-Claude BARTHELEMY, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France